CLINICAL TRIAL: NCT06806787
Title: Copeptin and Thirst: Possible Predictive Markers of Effectiveness of Bariatric Surgery?
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: COPTBAR
Record Dates: First submitted 2024-12-30; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective, non-pharmacological, spontaneous, single-center, interventional study.

DETAILED DESCRIPTION:
COPTBAR is a prospective, nonpharmacological spontaneous single-center interventional study.

Laboratory tests and imaging study (complete abdomen ultrasonography) for monitoring patients will be conducted in accordance with normal clinical practice. In addition, periodic copeptin assay will be performed. Each patient, within the study protocol, will be evaluated for 12 months; thereafter, each patient will fall under the follow-up visits provided by normal clinical practice and by Corporate Diagnostic Therapeutic Pathway (PDTA).

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 40 in the absence of comorbidities; BMI ≥ 35 associated with at least one comorbidity
* Age ≥ 18 and less than or equal to 65 years
* Written informed consent obtained

Exclusion Criteria:

Contraindications to bariatric surgery:

* severe psychiatric illness in the decompensation phase;
* drug or alcohol abuse;
* patient unwilling to follow periodic checkups and a dietary regimen pregnancy or lactation.

Factors that could alter ADH/copeptin:

* Obesity induced by other endocrinopathies or medications;
* Diabetes mellitus of any type;
* Malignant neoplasms or ongoing acute disease;
* Organ failure or chronic CNS and kidney disease;
* Hydro-electrolyte alterations;
* use of drugs that interfere with pituitary-adrenal axis, diuretics, anti-psychotics and psychopharmacological therapies, GLP1 receptor agonists, estro-progestin therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPTBAR is a prospective, nonpharmacological spontaneous single-center interventional study.
  Laboratory tests and imaging study (complete abdomen ultrasonography) for monitoring patients will be conducted in accordance with normal clinical practice. In addition, periodic copeptin assay will be performed. Each patient, within the study protocol, will be evaluated for 12 months; thereafter, each patient will fall under the follow-up visits provided by normal clinical practice and by Corporate Diagnostic Therapeutic Pathway (PDTA).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-03-14 (Estimated)

PRIMARY OUTCOMES:
Postoperative Weight Loss and Copeptin Concentration Association | through study completion, an average of 1 year
  To verify the existence of an association between postoperative weight loss and reduced copeptin concentration in patients with obesity undergoing laparoscopic sleeve gastrectomy surgery.
Correlation Between Copeptin Concentration and Thirst Perception | through study completion, an average of 1 year
  To verify the degree of correlation between copeptin concentration and thirst perception in patients with obesity undergoing laparoscopic sleeve gastrectomy surgery.

SECONDARY OUTCOMES:
Association Between Reduced Copeptin Concentration and Metabolic Parameters (Fasting Glucose, Insulin, HOMA-IR, Lipid Profile, HbA1c) in Patients Undergoing Laparoscopic Sleeve Gastrectomy | through study completion, an average of 1 year
  To verify, in patients with obesity undergoing laparoscopic sleeve gastrectomy surgery, the existence of an association between reduced copeptin concentration and improved metabolic parameters, assessed through fasting glucose, insulin levels, HOMA-IR index, lipid profile, and HbA1c measurements.
Correlation Between Thirst Perception (Assessed by a Validated Scale) and Metabolic Parameters (Fasting Glucose, Insulin, HOMA-IR, Lipid Profile, HbA1c) in Patients Undergoing Laparoscopic Sleeve Gastrectomy | through study completion, an average of 1 year
  To verify, in the same patients, the degree of correlation between thirst perception, evaluated using a validated thirst perception scale, and improvement of metabolic parameters, assessed through fasting glucose, insulin levels, HOMA-IR index, lipid profile, and HbA1c measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Uberto Pagotto, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy